CLINICAL TRIAL: NCT00183963
Title: A Pilot Clinical Trial to Evaluate the Biological Activity of Fulvestrant in Breast Ductal Carcinoma in Situ (DCIS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-03-7
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2012-12-06 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Fulvestrant

ARMS (4):
- 1 (No Intervention)
- 2 (Active Comparator): Tamoxifen 20 mg
  Interventions: Drug: Tamoxifen
- 3 (Active Comparator): Fulvestrant 250mg
  Interventions: Drug: Fulvestrant
- 4 (Active Comparator): Fulvestrant 500mg IM
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Tamoxifen — 20mg
  Arms: 2
Drug: Fulvestrant — 250mg
  Arms: 3
Drug: Fulvestrant — 500 mg IM
  Arms: 4

SUMMARY:
The subjects in this trial have been diagnosed as having a pre-cancerous disease of the breast called ductal carcinoma in situ (DCIS). This condition is associated with the development of breast cancer in up to 50% of cases.

The subjects are being asked to participate in this research study. They are being offered voluntary admission to this study to test the effects of a new investigational drug called Fulvestrant (Faslodex). This drug is approved by the United States Food and Drug Administration (FDA) for the treatment of advanced breast cancer but has not been approved for the treatment of DCIS. However, the FDA has given permission for the drug to be tested in this study. The purpose of this study is to find out if Fulvestrant has any effect on the subject's precancerous changes by comparing samples taken before and after receiving Fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with newly diagnosed DCIS. Women will be considered to be in menopause if they fall into one of the following groups:

  * Age > 60
  * Age > 45 with amenorrhea > 1 year with intact uterus
  * Status post bilateral oophorectomies
  * FSH/estradiol levels in postmenopausal range for the institution
* DCIS must have been diagnosed with a minimally invasive biopsy technique, such as a vacuum-assisted large core tool (Mammotome) or an equivalent method.
* There must be available tissue from the diagnostic biopsy to perform molecular markers.
* Baseline mammogram within 8 weeks of study entry.
* Serum creatinine less than or equal to 2.0 mg/dl.
* Total bilirubin less than or equal to 2.0 upper limit of normal (ULN), transaminases (SGOT and/or SGPT) and alkaline phosphatase may be up to 2.5 x institutional upper limit of normal (ULN), AGC greater than or equal to 1500, platelets greater than or equal to 100,000, Hemoglobin greater than or equal to 8.0 g/dl
* Peripheral neuropathy grade 0-1.
* No prior therapy for DCIS.
* SWOG performance status of less than or equal to 1
* All patients must provide informed written consent

Exclusion Criteria:

* Prior hormonal therapy (antiestrogens, estrogen, SERM's, progestins, or aromatase inhibitors) within 6 months of study entry.
* Underlying medical, psychiatric or social conditions that would preclude patient from receiving treatment.
* History of DVT or Pulmonary Embolism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Holmes, Principal Investigator — University of Southern California
Locations (1):
- Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the USC+LAC General Hospital between August 2006 to April 2008.
Pre-assignment Details: The study had no pre-assignment criteria.
Groups:
- Arm 1: Control Group: Placebo
- Arm 2: Tamoxifen Group: Tamoxifen 20 mg
  Tamoxifen : 20mg daily, by mouth x 21 days
- Arm 3: Low Dose Fulvestrant: Fulvestrant 250mg
  Fulvestrant : 250mg given on day 1, administered by IM Injection
- Arm 4: High Dose Fulvestrant: Fulvestrant 500mg
  Fulvestrant : 500mg given on day 1, administered by IM Injection
Period: Overall Study
Arm/Group | Arm 1: Control Group | Arm 2: Tamoxifen Group | Arm 3: Low Dose Fulvestrant | Arm 4: High Dose Fulvestrant
Started | 1 | 1 | 1 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Control Group | Arm 2: Tamoxifen Group | Arm 3: Low Dose Fulvestrant | Arm 4: High Dose Fulvestrant | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Molecular Changes in Markers of Cell Proliferation and Apoptosis Associated With Treatment
Description: Molecular measures of effect will be measured in tissue obtained at baseline biopsy (paraffin specimen) and on surgical specimen obtained at end of 3 weeks of treatment.
Time Frame: 6 months after treatment of last patient enrolled
Population: Analysis was not conducted since there was only 1 subject randomized on to each of the treatment arms.
Groups:
- Arm 2: Tamoxifen Group: 20 mg given by mouth daily for 21 days
- Arm 3: Low Dose Fulvestrant: 250 mg given on day 1, administered by IM Injection
- Arm 4: High Dose Fulvestrant: 500 mg given on day 1, administered by IM Injection
Arm/Group | Arm 1: Control Group | Arm 2: Tamoxifen Group | Arm 3: Low Dose Fulvestrant | Arm 4: High Dose Fulvestrant
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Changes in Mammographic Density
Description: The mammograms will be scanned and a validated computer based threshold method will be used to determine the mammographic densities.
Time Frame: 6 months after treatment of last patient enrolled
Population: Analysis was not conducted since there was only 1 subject accrued on to each of the treatment arms.
Arm/Group | Arm 1: Control Group | Arm 2: Tamoxifen Group | Arm 3: Low Dose Fulvestrant | Arm 4: High Dose Fulvestrant
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks after treatment
Arm/Group | Arm 1: Control Group | Arm 2: Tamoxifen Group | Arm 3: Low Dose Fulvestrant | Arm 4: High Dose Fulvestrant
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Control Group (N=1) | Arm 2: Tamoxifen Group (N=1) | Arm 3: Low Dose Fulvestrant (N=1) | Arm 4: High Dose Fulvestrant (N=1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction/extravasation changes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to insufficient accrual, analysis was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes